CLINICAL TRIAL: NCT06801860
Title: The Effectiveness of Chewing Gum for Reducing Cigarette Consumption and Promoting Smoking Cessation: A Pilot Randomized Controlled Trial
Brief Title: Chewing Gum for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Chew-to-Quit
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-01

CONDITIONS: Smoking Cessation
Keywords: Chewing gum; Behavioral intervention; Smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gum (Experimental): Participants in the intervention group will receive 1-2 packs of chewing gum over a 1-week intervention period. They will also receive a leaflet of usage tips for chewing gum, including 1) the potential benefits of chewing gum, 2) suitable usage time and dosage, and 3) the proper disposal of used gum.Additionally, participants in the intervention group will receive 2-week reminder message to boost gum usage.
  Interventions: Behavioral: Very brief smoking cessation advice; Behavioral: Chewing gum; Behavioral: Chewing gum usage leaflet; Behavioral: 2-week reminder message
- Unassisted quitting (Active Comparator): Participants in the unassisted quitting group (control group) will receive very brief smoking cessation advice (30 seconds) and a smoking cessation information booklet at baseline.
  Interventions: Behavioral: Very brief smoking cessation advice

INTERVENTIONS:
Behavioral: Very brief smoking cessation advice — All participants will receive very brief smoking cessation advice (guided by the AWARD model, assess, warning, refer, and do-it-again) with a smoking cessation information booklet onsite at baseline.
Behavioral: Chewing gum — Participants in the intervention group will receive 1-2 packs of chewing gum over a 1-week intervention period.
  Arms: Chewing gum
Behavioral: Chewing gum usage leaflet — A leaflet of usage tips for chewing gum, including 1) the potential benefits of chewing gum, 2) suitable usage time and dosage, and 3) the proper disposal of used gum.
  Arms: Chewing gum
Behavioral: 2-week reminder message — A 2-week reminder message guided by the Love and Care approach will be delivered to participants twice a week (a total of four).
  Arms: Chewing gum

SUMMARY:
The goal of this trial is to assess the feasibility, acceptability, and preliminary effectiveness of chewing gum to reduce cigarette consumption and promote smoking cessation. The main questions it aims to answer are: Do participants in the intervention group report a higher reduction in cigarette consumption, improved smoking cessation outcomes, and healthier oral health than the control group?

Researchers will compare chewing gum intervention to unassisted quitting to see if chewing gum works to cigarette reduction and smoking cessation.

Participants will:

1. Receive very brief smoking cessation advice and booklet at baseline.
2. Take chewing gum or unassisted quitting for 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. Residents of Hong Kong aged 18 or above
2. Smoking at least 1 cigarette per day over the past 3 months
3. Have the habit of chewing gum or are willing to use chewing gum
4. Participants who can communicate in Cantonese (including reading Chinese)
5. Expressing an intention to quit or reduce smoking
6. Capable of using instant messaging tools (e.g., WhatsApp, WeChat) for communication

Exclusion Criteria:

1. Having communication barriers (either physical or cognitive)
2. Currently participating in other smoking cessation programs or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Validated abstinence | 6-month follow-up
  Biochemically validated smoking abstinence will be measured by saliva cotinine level (exhaled carbon monoxide <4 ppm and salivary cotinine <30 ng/ml)

SECONDARY OUTCOMES:
Number of pieces used | 2-week, 3-month, and 6-month follow-ups
  The number of pieces used will be measured by a self-designed question: "On average, how many pieces of gum do you use every day?"
Frequency of use | 2-week, 3-month, and 6-month follow-ups
  The frequency of use will be measured by a self-designed question: "In the past seven days, how many days have you used chewing gum?"
Duration of use | 2-week, 3-month, and 6-month follow-ups
  Duration of use will be measured by a self-designed question: "How long do you typically use it at a time?"
Health effect | 2-week, 3-month, and 6-month follow-ups
  Health effect will be measured by a self-designed question: "Have you noticed any changes in your oral health after using chewing gum?"
The biochemically validated smoking abstinence | 6-month follow-up
  Smoking abstinence is defined by exhaled CO <4 ppm and salivary cotinine <30ng/ml
Self-reported 7-day point-prevalence abstinence | 2-week, 3-month, and 6-month
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up.
Self-reported smoking change | 2-week, 3-month, and 6-month follow-ups
  Self-reported change in number of cigarettes smoked daily of at least less 50% of the baseline number
Self-reported self-efficacy of quitting | 2-week, 3-month, and 6-month follow-ups
  Self-reported self-efficacy of quitting includes the perception of quitting importance, difficulty, and confidence, assessing by an item scaled with 0-10, respectively. The score of zero refers to very unimportant, very easy, or very unconfident. The score of 10 refers to very important, very difficult, or very confident, respectively. Higher score refers to higher perception of quitting importance, difficulty, and confidence.
Self-reported quit attempt | 2-week, 3-month, and 6-month follow-ups
  Self-reported quit attempt in the past 7 days.
Nicotine dependence level | 2-week, 3-month, and 6-month follow-ups
  The nicotine dependence level will be measured by the Fagerstrom Test for Nicotine Dependence (FTND). The score ranges from 0 to 10, with higher scores indicating greater nicotine dependence.
Smoking cessation services use | 2-week, 3-month, and 6-month follow-ups
  Using the smoking cessation service from hospitals or the government in Hong Kong
Self-reported intention to quit | 2-week, 3-month, and 6-month follow-ups
  Self-reported intention to quit in the next days

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Pokfulam, Hong Kong

IPD SHARING:
Plan to Share IPD: No